CLINICAL TRIAL: NCT00712361
Title: A Comparative Clinical Trial to Assess the Accuracy of the SoftTouch. A Novel Non-invasive Device for Measuring Peripheral Blood Glucose, Carbon Dioxide, pH, Hemoglobin, Hematocrit, SpO2, Peripheral Pulse and Blood Pressure.
Brief Title: A Comparative Study of the SoftTouch Non-Invasive Finger-Mounted Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cnoga Medical Ltd. (Industry)
Collaborators: Carmel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CM-CL-R-007; CMC 07015922 CMC 07015409 (Other: Carmel); HT 4502 (Other: helsinki Carmel); HTA 4502 (Other: Carmel)
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2009-12

CONDITIONS: Accuracy of the SofTouch Device Measuring Blood Glucose and Other Parameters
Keywords: Invasive; Non-Invasive; Peripheral blood parameters; Finger mounted device; Blood tissue; Tissue color distribution; Accuracy; Tissue pigmentation; pH; Hemoglobin; Hematocrit; SpO2; Blood pressure; Pulse; CO2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group A (Experimental): The group A incorporates three subgroups of individuals at various ages. A.1 Age: 16 - 30 A.2 Age: 31 - 60 A.3 Age > 60 All subgroups will be randomly distributed according to the following factors: BMI, gender, race and hematocrit.
  Interventions: Device: Non Invasive peripheral blood screening (Cnoga Medical Ltd.,SofTouch,OnlyTouch, CM-CL-R-007, CMC 07015922,HT 4502, HTA 4502)

INTERVENTIONS:
Device: Non Invasive peripheral blood screening (Cnoga Medical Ltd.,SofTouch,OnlyTouch, CM-CL-R-007, CMC 07015922,HT 4502, HTA 4502) — Non Invasive screening of various independent peripheral blood parameters: Glucose, hemoglobin, Hematocrit, blood pressure, pulse, SpO2, CO2, pH.
  Other Names: Cnoga Medical Ltd.; SoftTouch; SofTouch; Soft-Touch; OnlyTouch; CM-CL-R-007; CMC 07015922; HT 4502; HTA 4502

SUMMARY:
1. Aim:

   SoftTouch is a non-invasive device intending for use in the temporarily quantitative measurement of peripheral blood biomarkers. The aim of the clinical trial is to study the accuracy of the SoftTouch device compared with registered (FDA-approved) invasive and non-invasive devices.
2. Hypothesis:

Human physiological biomarkers may be measured from the color distribution of the internal or external (skin) tissue. The technology of the SoftTouch finger-mounted device is based on the color distribution of the peripheral blood tissue, which enables the measurement of certain biomarkers and vital signs under consideration.

DETAILED DESCRIPTION:
Description of the Method:

1. The method of measuring non-invasive peripheral physiological parameters such as Pulse, Blood Pressure, Blood pH, SpO2, CO2, Hemoglobin, Blood Glucose, Hematocrit and additional physiological parameters is based on the color distribution of a human tissue. SoftTouch is a finger-mounted device incorporated a dedicated light source and a color image sensor similar to a digital camera. The light transverses and is reflected from the tissue under consideration. Analyzing the tissue color distribution of the sampled real-time video in the frequency color space time domain may provide certain information about the biomarkers and vital-signs under consideration. The current study's goal is to find out if the results accuracy are satisfactory compared with regulatory cleared devices by the FDA and other notified bodies.
2. The Patient signals shall be recorded as is for algorithm improvement, future research of additional bio parameters and calibration.
3. the device is declared calibrated if executed successfully on the entire recorded data.
4. for non invasive blood glucose the device shall be provided to selected diabetic patients for the own use at home.

ELIGIBILITY:
INCLUSION CRITERIA:

Questions regarding INCLUSION must all be answered YES for subject study entry

1. Subject is 18 to 85 years of age? [ ]Yes
2. Finger skin surface to be tested is free of injury or skin disease? [ ]Yes
3. Subject is ambulatory? [ ]Yes
4. Subject is willing and able to comply with the study requirements? [ ]Yes
5. Subject is willing and able to provide written informed consent to participate in the study? [ ]Yes

   EXCLUSION CRITERIA:

   Questions regarding EXCLUSION must all be answered NO for subject study entry
6. Subject is currently hospitalized ambulatory free? [ ] No
7. Subject is currently abusing alcohol or illicit drugs, or has a history of alcohol abuse or illicit substance abuse within the preceding 2 years. For the purposes of the present study, alcohol abuse is arbitrarily defined as frequent consumption of alcoholic beverages with an average daily intake of more than 40gr of ethanol. Subject is currently on methadone maintenance treatment programs are NOT eligible for this study? [ ] No
8. Subject has a medical condition that requires frequent or prolonged use of systemic corticosteroids (eg. Severe asthma, severe arthritis or autoimmune conditions; organ transplantation, adrenal insufficiency)?[ ] No
9. The skin area to be tested clean of any damage (e.g. spotless, uncontaminated, dirt free, and hygienic)? [ ] No
10. Subject has any other concurrent medical or social condition likely to preclude compliance with the schedule of evaluations in the protocol, or likely to confound the efficacy or safety observations of the study (e.g. concurrent active malignancy; frequent or uncontrolled seizure disorder; severe psychiatric disorder requiring psychotropic medication; active tuberculosis, pneumonia or other severe infection under current treatment; lives in a country other than the investigative site; or has other medical or social circumstances likely to interfere with the schedule or evaluations? [ ] No
11. A history of treated malignancy that is not in complete remission of chemotherapy and/or radiotherapy and with additional surgical intervention during the preceding 3 years? [ ] No
12. Subject is enrolled or plans to enroll from this study for any personal reason ? [ ] No

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Non Invasive Screening of: Glucose, Hemoglobin, Hematocrit, Blood Pressure, Pulse, SpO2, CO2, pH. | up to 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Eli Zuckerman, Prof., Principal Investigator — Carmel Medical Center - Head of Liver Unit; Yosef Segman, PhD, Study Chair — Cnoga Medical Ltd.
Locations (4):
- Israel (4):
  - Patient's residence, Patient's Residence City, Patinet's Residence Province
  - Carmel Medical Center, Haifa
  - Lin Medical Center, Haifa
  - CNOGA Medical Ltd., Or Akiva

REFERENCES:
- [Background] References: 1. Indian J Med Res. 2007 Mar;125(3):275-96 2. Self-monitoring of blood glucose in diabetes. Drug Ther Bull. 2007 ;45(9):65-9. Blood glucose monitoring: reducing the cost, increasing the benefit. 4. Hussain F, Evans ND, Sachedina N, Pickup JC, In vivo glucose monitoring: the clinical reality and the promise. Biosens Bioelectron. 2005 Apr 15;20(10):1897-902. 5. Sims AJ, Menes JA, Bousfield DR, Reay CA, Murray A. Automated non-invasive blood pressure devices: are they suitable for use? Blood Press Monit. 2005 Oct;10(5):275-81. 6. Funahashi J, Ohkubo T, Fukunaga H, Kikuya M, Takada N, Asayama K, Metoki H, Obara T, Inoue R, Hashimoto J, Totsune K, Kobayashi M, Imai Y. The economic impact of the introduction of home blood pressure measurement for the diagnosis and treatment of hypertension. Blood Press Monit. 2005 Dec;10(6):307-10. 7. Bobrie G, Chatellier G, Genes N, Clerson P, Vaur L, Vaisse B, Menard J, Mallion JM. Cardiovascular prognosis of